CLINICAL TRIAL: NCT00280683
Title: Phase 2 Study: GCRC: Effects of L-arginine Supplementation on Exhaled Nitric Oxide and Clinical Exacerbations in Adults With Moderate to Severe Asthma
Brief Title: Effects of L-arginine Supplementation in Adults With Moderate to Severe Asthma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Center for Research Resources (NCRR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 200412788; UL1RR024146 (NIH); K30-04-Z001 (Other: UC Davis)
Record Dates: First submitted 2006-01-19; First posted 2006-01-23 (Estimated); Results first posted 2013-06-05 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Asthma
Keywords: Airway Inflammation; Moderate persistent asthma; Severe Persistent Asthma
MeSH Terms: conditions — Asthma | interventions — Arginine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arginine (Active Comparator): Enrolled subjects will take L-arginine orally, at 0.1 g/kg/day. Subjects will take three to four 1 g capsules (based on weight) of L-arginine twice daily for three months. L-arginine capsules were obtained from Jarrow Pharmaceuticals.
  Interventions: Drug: L-arginine
- Placebo (Placebo Comparator): Enrolled subjects took three to four placebo capsules that matched color and size of the intervention twice daily for three months. Matching placebo capsules were obtained from Jarrow Pharmaceuticals.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: L-arginine — subjects will take matching 0.01 g/kg/day of L-arginine in divided doses for thre months.
  Other Names: Arginine 1000
  Arms: Arginine
Drug: Placebo — Placebo tablets that match the L-arginine intervention tablets will be given for three months
  Other Names: Matching placebo tablets
  Arms: Placebo

SUMMARY:
Nitric oxide is an important marker of airway inflammation in asthma. Nitric oxide may have a protective role in patients with moderate to severe asthma. The investigators believe that a natural amino acid, L-arginine, that augments nitric oxide levels can decrease asthma exacerbations and improve the asthma care of moderate to severe asthma patients.

This study is a randomized, placebo controlled trial in which subjects will receive either 3 months of L-arginine supplementation or a placebo. The investigators will monitor subjects' symptoms, the number of asthma exacerbations, and lung function. In addition, we will draw blood, obtain induced sputum samples and measure exhaled breath nitric oxide levels at each monthly visit.

DETAILED DESCRIPTION:
The primary objective of this 3 month clinical study is to determine if supplemental L-arginine can decrease the number of asthma exacerbations in patients with severe asthma. L-arginine, a natural amino acid, produces nitric oxide (NO) when it is converted to L-citrulline in the presence of the nitric oxide synthase enzymes. We and others have found that NO can protect against allergic airway inflammation, airway hyperresponsiveness and airway fibrosis in various animal models. In addition, we have found that arginase I expression correlates strongly with the lymphocyte and eosinophil influx into the lung and this enzyme may regulate the airway inflammatory response. Our central hypothesis is that L-arginine will increase NO levels in the lung and decrease the number of acute exacerbations of asthma. It may do this by either decreasing the number of Th2 lymphocytes or down-regulating arginase I expression or both.

Our specific aims are, therefore,

1. To test the hypothesis, in a randomized, double-blinded, placebo controlled trial, that 3 months of L-arginine supplementation will decrease the number of acute asthma exacerbations in severe asthmatic patients,
2. To determine whether L-arginine decreases the ratio of peripheral blood Th2 to Th1 lymphocytes and
3. To determine whether L-arginine will modulate serum arginase I/II levels and their downstream products.

Patients will be recruited primarily from the UC Davis Asthma Network (UCAN) clinics, which focus on the care of severe asthmatics, and the study will be performed at the UC Davis/VA General Clinical Research Center.

ELIGIBILITY:
Inclusion Criteria:

* Moderate to severe persistent asthma
* Subject is stable on same asthma medications for at least one month
* If the subject is a woman of child-bearing age, a negative pregnancy test

Exclusion Criteria:

* Less than 18 yrs/ age
* Baseline Forced Expiratory Volume in 1 second (FEV1) <40% predicted
* Known or suspected allergy to L-arginine
* Pregnant women, nursing women, or women actively trying to achieve pregnancy
* Current smokers
* Subjects with more than a 15 pack-year history of smoking

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2004-12; Primary Completion 2008-11 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Kenyon, MD, Principal Investigator — University of California, Davis
Locations (1):
- University of California, Davis General Clinical Research Center, Sacramento, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between 2006-2008, moderate to severe persistent asthma patients, as defined by the NAEPP Expert Panel Reports, were eligible for enrollment [10]. Most subjects were recruited from the UC Davis Asthma Network clinics, which are referral clinics for patients with difficult to control asthma.
Pre-assignment Details: The randomization process and disbursement of L-arginine (0.05 g/kg twice daily; 6-10 g/day) and placebo were done by the UC Davis Investigational Drug Service.Eligible subjects had documented moderate to severe persistent asthma, were at least 18 years of age, not pregnant, and able to give consent.
Groups:
- Arginine; Placebo: 2.3. L-Arginine Intervention The randomization process and disbursement of L-arginine and placebo were done by the UC Davis Investigational Drug Service to ensure that both the physician and participant were blinded.
Period: Overall Study
Arm/Group | Arginine | Placebo
Started | 10 | 10
Completed | 8 (Reasons for subjects discontinuing included inability to adhere to the schedule or adverse event.) | 7
Not Completed | 2 | 3
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Adverse Event | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Arginine: 2.3. L-Arginine Intervention The randomization process and disbursement of L-arginine (0.05 g/kg twice daily; 6-10 g/day) and placebo were done by the UC Davis Investigational Drug Service to ensure that both the physician and participant were blinded. The subjects began the study medication on day 0 and continued for 90 days and were asked to discontinue use of any nutritional supplements prior to the start of the study.
- Placebo: Placebo intervention
- Total: Total of all reporting groups
Arm/Group | Arginine | Placebo | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9 | 9 | 18
  >=65 years | 1 | 1 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.1 (15.4) | 50.8 (15.1) | 52.0 (15.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 8 | 16
  Male | 2 | 2 | 4
FEV1 Percent Predicted [Mean (Standard Deviation); unit: Percent] | 75 (17.5) | 70.8 (18.5) | 72.9 (18.0)
Exhaled Nitric oxide [Mean (Standard Deviation); unit: ppb (parts per billion)] — The secondary clinical endpoints that were measured included the patient symptom diary, daily short acting β-agonist use, St. George's Respiratory questionnaire, daily PEF diary, forced expiratory volume in one second (FEV1), and forced expiratory volume in one second to forced vital capacity ratio (FEV1/FVC) measurements performed at the monthly visits, exhaled NO concentration and induced sputum eosinophil percent counts
  ppb (parts per billion) | 28.2 (16.4) | 24.4 (17.6) | 26.3 (17)

OUTCOME MEASURES:

1. Primary Outcome: Number of Asthma Exacerbations in Three Months
Description: Asthma exacerbation is a composite endpoint. An asthma exacerbation is defined as any of the following: a) a drop in the morning peak expiratory flow rate (PEF) >30% from baseline on 2 consecutive days, b) a need for initiation of or increased dose of inhaled corticosteroids, or the c) doubling of short-acting rescue β-agonist drug use (e.g.Albuterol) on two consecutive days. Any one of these three counts as one asthma exacerbation.
Time Frame: 3 months
Population: Our original power analysis was based on an expected minor exacerbation rate of 3-4 per month.
Measure: Number; unit: exacerbations
Groups:
- Arginine: The L-arginine 1g tablets were from Jarrow formulas (Los Angeles, CA). The name of these tablets is Arginine 1000.
- Placebo: Matching placebo tablets were made by Jarrow Formulas.
Arm/Group | Arginine | Placebo
Number analyzed (Participants) | 10 | 10
exacerbations | 30 | 31

2. Secondary Outcome: L-arginine Serum Concentration
Time Frame: 90 days
Measure: Mean (Standard Error); unit: pmol/100ul
Groups:
- Arginine: L-Arginine Intervention The randomization process and disbursement of L-arginine (0.05 g/kg twice daily; 6-10 g/day) and placebo were done by the UC Davis Investigational Drug Service to ensure that both the physician and participant were blinded. The subjects began the study medication on day 0 and continued for 90 days and were asked to discontinue use of any nutritional supplements prior to the start of the study.
- Placebo: Matching placebo tablets were disbursed by the Investigational Drug Service.
Arm/Group | Arginine | Placebo
Number analyzed (Participants) | 10 | 10
pmol/100ul | 0.002 (0.0006) | 0.0011 (0.0002)

ADVERSE EVENTS:
Time Frame: 1 year intervals
Groups:
- Arginine: L-arginine 1 g tablets were made by Jarrow Formulas.
- Placebo: Matching placebo tablets were purchased from Jarrow Formulas.
Arm/Group | Arginine | Placebo
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 1/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arginine (N=10) | Placebo (N=10)
Hypertension (Cardiac disorders) | 0 (0) | 1 (1) — One subject in the placebo group was unblinded from the study and discontinued from study drug because of an increased in blood pressure. Blood pressure returned to normal.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No